CLINICAL TRIAL: NCT07207317
Title: Laparoscopic Ileocecal Reconstruction Right Hemicolectomy (LIRRH) Trial for the Right-sided Colon Cancer
Brief Title: LIRRH Trial for the Right-sided Colon Cancer
Acronym: LIRRH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chaoxi Zhou (Other)
Responsible Party: Sponsor-Investigator, Chaoxi Zhou, Associate Chief Physician, Department of General Surgery, Hebei Medical University Fourth Hospital
Organization: Hebei Medical University Fourth Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KS060; 2025KS060 (Other: Ethics Committee of the Fourth Hospital of Hebei Medical University)
Record Dates: First submitted 2025-09-15; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Ascending Colon Cancer; Proximal Transverse Colon Cancer
Keywords: Right-sided colon cancer; Laparoscopic right hemicolectomy; Ileocecal reconstruction; Randomized controlled trial; Disease-free survival; TRH; LIRRH

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to either the LIRRH arm or the TRH arm and followed in parallel until completion of the trial; no crossover or factorial design is employed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIRRH group (Experimental): Participants will undergo laparoscopic ileocecal-reconstruction right hemicolectomy (LIRRH), in which the ileocecal junction is reconstructed; procedure follows the same oncologic resection margins as standard laparoscopic surgery.
  Interventions: Procedure: Laparoscopic ileocecal-reconstruction right hemicolectomy (LIRRH)
- TRH group (Active Comparator): Participants will undergo traditional laparoscopic right hemicolectomy (TRH) with standard en-bloc mesenteric resection and ileocolic anastomosis
  Interventions: Procedure: traditional laparoscopic right hemicolectomy (TRH)

INTERVENTIONS:
Procedure: Laparoscopic ileocecal-reconstruction right hemicolectomy (LIRRH) — The ileocolic vessels are divided at their roots, and lymph nodes of stations 203, 202, and 201 are dissected. The right colic and middle colic vessels are also divided at their roots, and the surrounding lymphatic and adipose tissue (stations 211/212/213 and 221/222/223) is cleared. The transverse colon is transected 10 cm distal to the tumor, and the ileum is divided 10 cm proximal to the ileocecal region. After tailoring the ileal mesentery, an end-to-end ileo-transverse colonic anastomosis is performed. Using a seromuscular suture, the ileum and its tailored mesentery are invaginated into the wall of the transverse colon 2 cm proximal to the anastomosis, thereby reconstructing the ileocecal valve complex.
  Arms: LIRRH group
Procedure: traditional laparoscopic right hemicolectomy (TRH) — The ileocolic vessels are divided at their roots, and lymph nodes of stations 203, 202, and 201 are dissected. The right colic and middle colic vessels are likewise divided at their roots, and the surrounding lymphatic and adipose tissue (stations 211/212/213 and 221/222/223) is cleared. The transverse colon is transected 10 cm distal to the tumor, and the ileum is divided 10 cm proximal to the ileocecal junction. An end-to-side or side-to-side ileo-transverse colonic anastomosis is then performed.
  Arms: TRH group

SUMMARY:
The aim of this clinical trial is to compare the short- and long-term outcomes of laparoscopic ileocecal reconstruction right hemicolectomy (LIRRH) with those of traditional laparoscopic right hemicolectomy (TRH) for ascending and proximal transverse colon cancer.

DETAILED DESCRIPTION:
This is a prospective, single-center, open-label, randomized controlled clinical trial. Eligible patients will be randomly assigned (1:1) to undergo either LIRRH or TRH and will receive the corresponding surgical procedure.

Primary endpoint: 3-year disease-free survival (DFS).

Secondary endpoints:

1. Complications within 90 days postoperatively;
2. Pathology-related indicators, including positive margin rate, number of harvested lymph nodes, and lymph-node metastasis rate;
3. Assessment of postoperative intestinal microbiota changes;
4. 5-year overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* ASA physical status ≤ III
* Endoscopy and biopsy-proven colon adenocarcinoma
* Contrast-enhanced abdominal CT showing primary tumor located in the ascending colon or proximal transverse colon (proximal one-third)
* Pre-operative clinical stage: TanyNanyM0
* Able to understand the study protocol, willing to participate, and provide written informed consent

Exclusion Criteria:

* History of hypertensive crisis or hypertensive encephalopathy.
* Severe cardiopulmonary insufficiency or any other contraindication to surgery.
* Uncorrectable electrolyte disturbances (e.g., potassium, calcium, magnesium).
* Evidence of significant bleeding diathesis or high hemorrhagic risk:
* Prior intracranial or intraspinal hemorrhage.
* Tumor invading major vessels with obvious bleeding risk.
* Thrombotic or embolic event within 6 months before study treatment, or significant vascular disease (e.g., surgical-repair aortic aneurysm).
* Clinically relevant hemoptysis or tumor bleeding of any cause within 1 month before screening.
* Therapeutic-dose anticoagulation within 2 weeks before study treatment (except low-molecular-weight heparin).
* Antiplatelet therapy within 10 days before study treatment (e.g., aspirin > 325 mg/day, clopidogrel > 75 mg/day, dipyridamole, ticlopidine, cilostazol).
* Active tuberculosis.
* Any active autoimmune disease or history of autoimmune disease with expected recurrence (including but not limited to SLE, RA, autoimmune hepatitis, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyper- or hypothyroidism, asthma requiring bronchodilators).
* Pre-operative evidence of synchronous multiple primary colorectal cancers or other conditions requiring additional bowel resection.
* Pre-operative imaging or intra-operative findings showing:
* Tumor infiltration into adjacent organs requiring multi-visceral resection;
* Distant metastasis;
* Unresectable (unable to achieve R0) disease.
* Other malignancies within the past 5 years, or familial adenomatous polyposis; except cured carcinoma in situ of the cervix, basal-cell carcinoma, papillary thyroid carcinoma, or cutaneous squamous-cell carcinoma.
* Intestinal obstruction, perforation, or bleeding requiring emergency surgery.
* Patient unsuitable or unable to tolerate laparoscopic surgery.
* Pregnant or lactating women.
* History of psychiatric disorders precluding compliance.
* Prior neoadjuvant therapy.
* Multidisciplinary team (MDT) decision that the patient is not appropriate for the study.
* Patient unable to understand the study conditions/objectives and refuses to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival (DFS) | From date of randomization until the date of first documented recurrence or death from any cause, assessed up to 36 months
  DFS is defined as the time from randomization to the earliest date of locoregional recurrence, distant metastasis, second primary colorectal cancer, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
10-day postoperative diarrhea rate | Within 10 days after surgery
  The proportion of patients experiencing diarrhea within 10 days after surgery, graded by the Clavien-Dindo classification system.
  Unit of Measure: %
15-day postoperative ileus rate | 15 days after surgery
  The proportion of patients experiencing ileus within 15 days after surgery, graded by the Clavien-Dindo classification system.
  Unit of Measure: %
Pathology-related composite indicator | Immediate (on specimen examination, within 7 days post-op)
  A composite indicator related to pathology, including the positive margin rate, the number of harvested lymph nodes, and the lymph node metastasis rate. These indicators will be aggregated into a single reported value through a composite score or statistical analysis.
  Unit of Measure: Composite score or percentage (%)
Postoperative gut microbiota diversity | 6 months and 1 year post-surgery
  The diversity of gut microbiota assessed by 16S rRNA gene sequencing at 6 months and 1 year post-surgery. The primary metrics include the Shannon diversity index and the Chao1 richness index.
  Unit of Measure: Shannon diversity index (dimensionless) and Chao1 richness index (number of OTUs)
5-year overall survival | From randomization to death from any cause, assessed up to 60 months
  Overall survival (OS) is defined as the time from randomization to death from any cause; survivors will be censored at the last follow-up. Unit of Measure: %

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified individual participant data will be shared: baseline demographics, operative variables, pathologic staging, adjuvant therapy details, recurrence and survival outcomes, and serious adverse events. Data will be provided in CSV format with a data dictionary and variable coding manual.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after primary publication (est. Q4 2027) through 2032 (5 years from sharing).
Access Criteria: De-identified IPD, along with the protocol, SAP, and analytic code, will be made available to qualified researchers who provide a methodologically sound proposal, IRB/ethics approval documentation, and a signed data-access agreement. Data will be accessed through a secure, password-protected academic repository (e.g., Zenodo) after approval by the study steering committee.
URL: https://pending.org